CLINICAL TRIAL: NCT05520151
Title: Influence of Preoperative Immunomodulation by Oral Impact® on Postoperative Complications Following Cystectomies and Nephrectomies
Brief Title: Influence of Preoperative Immunomodulation by Oral Impact on Postoperative Complications Following Cystectomies & Nephrectomies
Acronym: IMPACTURO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Robert Ballanger (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GHT-CHIRB -20220411
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Urological Manifestations
Keywords: cystectomy,; nephrectomy,; laparotomies; reduction of postoperative complications
MeSH Terms: conditions — Urological Manifestations | interventions — Organization and Administration

STUDY DESIGN:
Intervention Model Description: Multicentric, prospective non-randomized clinical study comparing the group of patients who received a 7-days course of ORAL IMAPCT to a retrospective cohort of patients operated between 2016 and 2019: cystectomy and nephrectomy by laparotomy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ORAL impact group (Experimental): This group of patients will receive a 7-days course of IMPACT ORAL 20 days before the surgery
  Interventions: Dietary Supplement: ORAL IMPACT treatment
- control (Other): a retrospective cohort of patients operated between 2016 and 2019 by nephrectomy cystectomy and laparotomy who did not receive oral impact
  Interventions: Other: control

INTERVENTIONS:
Dietary Supplement: ORAL IMPACT treatment — the group of patients will be received a 7-days course of ORAL IMPACT
  Other Names: Monitoring of postoperative albumin on days 1, 3, 5, 7, and 10; correction of postoperative hypoalbuminemia (<35 g/L) by albumine 20% administration in case of postoperative complications
  Arms: ORAL impact group
Other: control — no intervention
  Arms: control

SUMMARY:
any studies have shown the benefit of perioperative Oral Impact immunomodulation in gastrointestinal, ENT, gynecological and cardiac surgery. Studies in major Urological surgery are rare and not very contributory. The expected benefit is a reduction in postoperative complications and the average length of stay.

DETAILED DESCRIPTION:
Major surgery induces traumatic stress due to the surgical aggression which could lead to major postoperative complications and death when the patient organism is not ready or prepared to support this intense stress. Malnutrition can be caused by chronic starvation, chronic inflammatory disease and acute injury (stress, acute inflammation). Therefore, nutritional supplements are indicated for patients who do not meet their energy needs through oral food ingestion. Immune-modulating nutrient-enriched products containing arginine, Omega-3 polyunsaturated fatty acids (PUFAs), nucleic acids, vitamins and antioxidants (selenium) like ORAL IMPACT (Nestlé) can modulate immune and inflammatory processes in burn, trauma, major surgery and improving clinical outcomes. These immune-modulating nutrient-enriched products have shown their ability to decrease postoperative complications up to 50% in patients undergoing non-gastrointestinal major surgery and length of hospital and ICU stay (Jie B 2012, Drover 2011). Mortality benefits have been demonstrated in one study focused on Neck and Head surgery. (Buijs N, 2010) Before 2019, in our urology surgery setting, it seemed that the postoperative complications rate was clinically increasing despite reliable surgeons and excellent surgery techniques and procedures. It appeared that the sources of these complications might be the weakness of the patients against major surgical stress. Patients might have been malnourished. The nutritional status had been omitted from our preoperative anesthesia assessment and no perioperative nutritional rehabilitation had been performed.

The effect of immune-modulating nutrient-enriched products had been demonstrated mostly in gastrointestinal surgery but also in non-gastrointestinal surgeries such as neck and head cancer surgery, gynecologic cancer surgery and cardiac surgery. There are not studies conducted in urologic major surgery.

Reducing the number of post-operative complications is a major challenge in surgery because they cause an increase in the length of stay, which translates into higher hospital costs for the community. Surgery generates major metabolic stress that the human body must manage. This metabolic stress will manifest itself in an increase in catabolism and a decrease in anabolism, resulting in protein-energy malnutrition in the patient if they are insufficiently prepared. Preoperative undernutrition is one of the risk factors for major postoperative complications.

Moreover, postoperative infection can occur despite the Oral Impact treatment and associated iron and protein-caloric rehabilitation. It is linked to postoperative hypoalbuminemia. The antimicrobial role of albumin in the body is significant due to its antioxidant power. Reduced, non-oxidized albumin is the primary antioxidant in the body. Postoperative inflammation consumes reduced albumin, thereby diminishing the body's antioxidant capacity and exposing it to complications and nosocomial infections. The exogenous supply of reduced albumin is therefore indispensable. The liver's albumin synthesis yield is too low in this inflammatory context, amounting to approximately one vial of 20% albumin per day. Preoperatively, the correction of any hypoalbuminemia is anticipated through the nutritional rehabilitation implemented with the dietitian team. The timing of the surgery does not always allow the body to correct this hypoalbuminemia on its own. It is also essential to correct it postoperatively, in case of complications if necessary, through the exogenous supply of 20% reduced albumin.

Numerous studies have shown the benefit of perioperative Oral Impact immunomodulation in gastrointestinal surgery, ear, nose and throat surgery, gynecological and cardiac surgery.

No studies have been done in major Urological surgery The proposed study will be the first formal evaluation of the benefits and risks of using ORAL IMPACT in the preoperative period of urological surgery. The choice of this clinical project for this research question is justified by the proven benefit of this food substitute perioperatively in gastrointestinal, ear, nose and throat, gynecological and cardiac surgery. We hypothesize that Oral Impact will protect against major postoperative complications and prolonged hospital stay for patients undergoing urological surgery. There are no current guidelines recommending or discouraging the prescription of ORAL IMPACT in urological surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Scheduled major urological surgery: scheduled: cystectomy, nephrectomy, other laparotomies.
* Having expressed their free and informed consent.
* Affiliated to a social security scheme

Exclusion Criteria:

* Immune deficiency.

  * HIV infection.
  * Curative surgery for chronic urinary tract infection.
  * Urgent surgery.
  * Inability to take oral impact 7 days before surgery.
  * Unstable psychiatric state.
  * Infection with COVID 19 during postoperative stay.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Rate of major postoperative complications | 3 months
  the number of postoperative complications during this study for each patient

SECONDARY OUTCOMES:
Length of stay in hospital (LOS). | 3 months
  Length of stay in hospital (LOS). durind the participation of each patient
Number of admissions in intensive care setting for severe complications. | 3 months
  Number of admissions in intensive care setting for severe complications after major urological surgery.
Rate of transfusions of red blood cells. | 3 months
  Rate of transfusions of red blood cellsduring hospitalisation and after major urological surgery.
mortality rate | 3 months
  3-month mortality rate
Incidence of postoperative hypoalbuminemia | 10 days post-surgery
  albumin analysis
the average rate of postoperative hypoalbuminemia | 10 days post-surgery
  albumin analysis

CONTACTS AND LOCATIONS:
Overall Officials: Serge NDOKO, MD, Principal Investigator — Robert ballanger; MAtthieu CAMBY, MD, Principal Investigator — Centre Hospitalier Intercommunal André Grégoire
Locations (2):
- France (2):
  - CHI Robert Ballanger, Aulnay-sous-Bois
  - CHI André Grégoire, Montreuil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Finnerty CC, Mabvuure NT, Ali A, Kozar RA, Herndon DN. The surgically induced stress response. JPEN J Parenter Enteral Nutr. 2013 Sep;37(5 Suppl):21S-9S. doi: 10.1177/0148607113496117. PMID 24009246
- [Result] Katona P, Katona-Apte J. The interaction between nutrition and infection. Clin Infect Dis. 2008 May 15;46(10):1582-8. doi: 10.1086/587658. PMID 18419494
- [Result] Argiles JM. Cancer-associated malnutrition. Eur J Oncol Nurs. 2005;9 Suppl 2:S39-50. doi: 10.1016/j.ejon.2005.09.006. PMID 16437757
- [Result] Barker LA, Gout BS, Crowe TC. Hospital malnutrition: prevalence, identification and impact on patients and the healthcare system. Int J Environ Res Public Health. 2011 Feb;8(2):514-27. doi: 10.3390/ijerph8020514. Epub 2011 Feb 16. PMID 21556200